CLINICAL TRIAL: NCT04980001
Title: Trauma Informed Childhood Obesity Care for Low-Income Minorities in Primary Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was not started due to several factors: partial IRB approval; limited community partner engagement; and grant funding support expired.
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Principal Investigator, Angela Venegas, Assistant Professor, Charles Drew University of Medicine and Science
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1766233-1
Record Dates: First submitted 2021-07-08; First posted 2021-07-28 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Childhood Obesity
Keywords: trauma informed care
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: All participants will have access to the FOCUS TIC-COM intervention. The health care providers at the family medicine clinic within MLK-OPC will be trained to implement FOCUS TIC-COM with children who are overweight or obese. The investigators plan to survey and perform focus groups with health care providers and the parents / caregivers of children who were identified as overweight or obese by their doctor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOCUS TIC-COM arm (Experimental): Health care providers will be trained in FOCUS TIC-COM through professional development and from this group the investigators plan to recruit participants for the surveys about the training, intervention feasibility and acceptability. Health care providers will be encouraged to implement FOCUS TIC-COM will all of their pediatric patients who are overweight/obese.
  Parents / Caregivers of children who are overweight or obese will be recruited into the study after exposure to the intervention. Only those exposed to the intervention will be recruited to participate in the study which includes one survey and focus groups.
  Interventions: Behavioral: Families OverComing Under Stress Trauma Informed Care in Childhood Obesity among Minorities (FOCUS TIC-COM)

INTERVENTIONS:
Behavioral: Families OverComing Under Stress Trauma Informed Care in Childhood Obesity among Minorities (FOCUS TIC-COM) — FOCUS TIC-COM is a program that helps doctors coach families to recognize how emotions or feelings about various life stressors may affect a child's dietary choices and physical activity. FOCUS TIC-COM is for families of children who have been identified by their doctor as overweight or obese. The goal of the program is to help children and their families understand how their mental health may impact their physical health and develop strategies to address their mental health needs.

SUMMARY:
The purpose of this pilot study is to examine changes in childhood obesity associated with the implementation of a Trauma Informed Care approach with weight counseling and management among low-income minority children in a primary care setting.

DETAILED DESCRIPTION:
Prospective mixed methods pilot study, using both qualitative and quantitative measures. This study will be conducted in two phases. In Phase 1 (Year 1), the investigators plan to use a modified Delphi procedure called the RAND/UCLA Appropriateness Method in which the investigators will form a multidisciplinary panel to develop a consensus of incorporating the TIC practices based on FOCUS into current best practices for childhood obesity prevention and treatment among low-income minorities to be facilitated by primary care providers. In Phase 2 (Year 2), the investigators will train and implement the Primary Care Provider-mediated FOCUS TIC-COM among providers for obese children and their caregivers / parents in the MLK OPC Family Medicine Clinic. During this phase, the investigators plan to examine the feasibility and acceptability of delivering the FOCUS TIC-COM in the primary care setting at MLKOPC through surveys and focus groups with both providers and the parents / caregivers of overweight / obese children. The investigators will also explore whether the FOCUS TIC-COM impact on childhood obesity (as perceived by child's parent / caregiver) and increase linkages to behavioral health care regarding trauma / toxic stress. At 3 month intervals, the investigators will train a subset of providers in the intervention and they will implement the intervention immediately after training.

ELIGIBILITY:
Year 1:

Inclusion Criteria:

• Adult Experts (>18 years old) in the fields of trauma informed care and childhood obesity among low-income minorities

Exclusion Criteria:

• Individuals outside of the fields of trauma informed care or childhood obesity

Year 2:

Inclusion Criteria:

* Parents / Caregivers of overweight/obese children (ages 2-17 years old) in MLK-OPC who speak English or Spanish
* Primary Care Providers (>18 years old) who work in the Family Medicine Clinic of the MLK-OPC

Exclusion Criteria:

* Parents / Caregivers of children that are not overweight/obese and/or under 2 years old
* Parent or caregiver that speaks a language other than English or Spanish
* Primary Care Providers who do not work in the Family Medicine Clinic of the MLK-OPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
RAND/UCLA Appropriateness Method - Expert Panel Ratings / Consensus | Four rounds of rating over the course of 6 month to 1 year (Year 1 of study)
  The investigators plan to use a modified Delphi procedure called the RAND/UCLA Appropriateness Method to reach consensus regarding the content and implementation of a Primary Care Provider-mediated FOCUS TIC-COM approach to address childhood obesity in low-income minority communities. The RAND/UCLA Appropriateness Method consists of four rounds of rating clinical indicators or practice guidelines derived from current literature on TIC that will be incorporated into the current standard of childhood obesity prevention and management. A benefit-to-cost ratio will be rated on a 9 point Likert scale, where 1 means that the expected harms greatly outweigh the expected benefits in relation to cost, and 9 means that the expected benefits greatly outweigh the expected harms in relation to cost. Necessity rating scale will be on a Likert scale of 1 to 9, where 1 means that the practice guideline is not necessary at all, and 9 means that the practice guideline is extremely necessary.
FOCUS TIC-COM Training Evaluation - Provider's Perceived confidence | Baseline and immediately after training (Year 2 of study)
  The investigators plan to conduct a pre/post training evaluation measuring perceived confidence in FOCUS TIC-COM approach for overweight/obese children. The investigators will use a 5 point likert scale to measure confidence level in FOCUS TIC-COM approach, where 1 means "not confident at all" and 5 means "very confident". The 5 point likert scale for confidence has the following values: 1 means "not confident at all"; 2 means "not very confident"; 3 means "somewhat confident"; 4 means "fairly confident"; and 5 means "very confident".
Health care provider satisfaction of FOCUS TIC-COM | Last 6 months of Year 2 of study
  The investigators plan to collect health care provider satisfaction in delivering the FOCUS TIC-COM. The investigators will measure satisfaction of various elements of the intervention using a 5 point Satisfaction Likert scale, where 1 means "very unsatisfied" and 5 means "very satisfied".
Parent / Caregiver satisfaction of FOCUS TIC-COM | Last 6 months of Year 2 of study
  The investigators plan to collect parent / caregiver satisfaction in receiving the FOCUS TIC-COM intervention. The investigators will measure satisfaction of various elements of the intervention using a 5 point Satisfaction Likert scale, where 1 means "very unsatisfied" and 5 means "very satisfied".
Feasibility and acceptability of delivering FOCUS TIC-COM in the primary care setting, as perceived by caregivers/parents of low-income minority obese children and their providers | Last 6 months of Year 2 of study
  The investigators will conduct focus groups with both health care providers and parents/caregivers of overweight/obese children exposed to FOCUS TIC-COM to assess intervention feasibility and acceptability. The investigators will ask questions in the focus group discussion on whether the Primary Care Provider-mediated FOCUS TIC-COM is relevant, appropriate and sustainable for the primary care setting and if the intervention should be disseminated. In addition, the investigators will examine the demand, practicality, adaptation, integration, expansion and efficacy of the intervention through the focus group discussion. The focus group questions will be derived from the RE-AIM framework: Reach into the target population; Effectiveness / Efficacy; Adaptation by target settings, institutions, and staff; Implementation - consistency and cost of delivery; Maintenance of intervention effects.

SECONDARY OUTCOMES:
Calculated child BMI per parent / caregiver report | Last 6 months of Year 2 of study
  The investigators plan to collect parent / caregiver reported height (in meters squared) and weight (kilograms) of their child who received the FOCUS TIC-COM intervention. The height and weight of the child will be aggregated to calculate the child's body mass index (BMI).
Parent-reported linkages to behavioral health services | Last 6 months of Year 2 of study
  The investigators will ask parents / caregivers if their child who is overweight / obese was referred to behavioral health services by their health care provider. The investigators will also ask if those services were obtained or not.

CONTACTS AND LOCATIONS:
Overall Officials: Angela L Venegas-Murillo, MD MPH MS, Principal Investigator — Charles Drew University of Medicine and Science

IPD SHARING:
Plan to Share IPD: No